CLINICAL TRIAL: NCT02423317
Title: A Comparative Evaluation of Airtraq Optical LaryngoscopeTM and Miller Blade in Pediatric Patients Undergoing Elective Surgery Requiring Tracheal Intubation.
Brief Title: Comparison of Miller's Blade and Airtraq Laryngoscope in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Bikramjit Das, Assistant Professor, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DN 182/FM
Record Dates: First submitted 2015-03-29; First posted 2015-04-22 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Intubation, Intratracheal
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation with Miller's blade (Active Comparator): After induction and muscle paralysis, Miller's blade was introduced in the patient's mouth. After visualization of vocal cord, patient was intubated with appropriate sized tracheal tube.
  Interventions: Device: Intubation with Miller's blade
- Intubation with Airtraq laryngoscope (Experimental): After induction and muscle paralysis, Airtraq laryngoscope's blade was introduced in the patient's mouth. After visualization of vocal cord as a reflected image in the viewfinder of the device, patient was intubated with appropriate sized tracheal tube.
  Interventions: Device: Intubation with Airtraq

INTERVENTIONS:
Device: Intubation with Miller's blade — Intubation is insertion of a hollow tube inside the trachea. It is done after laryngoscopy with Miller's blade.
  Arms: Intubation with Miller's blade
Device: Intubation with Airtraq — Intubation is insertion of a hollow tube inside the trachea. It is done after laryngoscopy with Airtraq.
  Arms: Intubation with Airtraq laryngoscope

SUMMARY:
The Airtraq optical laryngoscope has recently been available in pediatric sizes. The investigators compared the efficacy of Airtraq with the Miller laryngoscope as intubation devices in paediatric patients. This prospective, randomized study was conducted in a tertiary care teaching hospital. Sixty American Society of Anesthesiologists (ASA) grade I-II paediatric patients of 2-10 years, posted for routine surgery requiring tracheal intubation were randomly allocated to undergo intubation using a Miller (n = 30) or Airtraq (n = 30) laryngoscope. The primary outcome measures were time of intubation, ease of intubation, number of attempts and POGO score. We also measured hemodynamic changes and airway trauma.

DETAILED DESCRIPTION:
After approval from the institutional Ethical Committee, 60 patients were studied. A randomised prospective study was planned to compare size 1 Airtraq (Prodol Meditec S.A., Vizcaya, Spain) with Miller blade of same size.

The children included in the study were 2-10 years of age, American Society of Anesthesiologists (ASA) physical status I-II and posted for elective surgeries requiring tracheal intubation. The following were excluded from the study: (i) patients with upper respiratory tract symptoms, (ii) those at risk of gastroesophageal regurgitation and (iii) those with airway-related conditions such a trismus, limited mouth opening, trauma or mass. Sixty patients were equally randomized to one of the two groups (Airtraq and Miller) of 30 each for airway management using a computer-generated randomization program.

Written informed consent was taken from the parents prior to intervention and a standardized protocol for anesthesia was maintained for all cases. All the children were kept nil per mouth as per standard guidelines. Intubation attempts were taken using Airtraq or Miller on a random basis.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists physical status I-II,
2. elective surgeries requiring tracheal intubation

Exclusion Criteria:

1. patients with upper respiratory tract symptoms,
2. those at risk of gastroesophageal regurgitation and
3. those with airway-related conditions such a trismus, limited mouth opening, trauma or mass.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahin N Jamil, M.D., Study Director — J.N.Medical College, Aligarh Muslim University

REFERENCES:
- [Background] Maharaj CH, Higgins BD, Harte BH, Laffey JG. Evaluation of intubation using the Airtraq or Macintosh laryngoscope by anaesthetists in easy and simulated difficult laryngoscopy--a manikin study. Anaesthesia. 2006 May;61(5):469-77. doi: 10.1111/j.1365-2044.2006.04547.x. PMID 16674623
- [Background] Sorensen MK, Holm-Knudsen R. Endotracheal intubation with airtraq(R) versus storz(R) videolaryngoscope in children younger than two years - a randomized pilot-study. BMC Anesthesiol. 2012 Apr 30;12:7. doi: 10.1186/1471-2253-12-7. PMID 22545575
- [Background] White MC, Marsh CJ, Beringer RM, Nolan JA, Choi AY, Medlock KE, Mason DG. A randomised, controlled trial comparing the Airtraq optical laryngoscope with conventional laryngoscopy in infants and children. Anaesthesia. 2012 Mar;67(3):226-31. doi: 10.1111/j.1365-2044.2011.06978.x. PMID 22321076
- See also: Official web site of Airtraq optical laryngoscope — http://www.airtraq.com/index.php?option=com_content&task=view&id=200&Itemid=329.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.4 (1.78) | 6.15 (2.64) | 5.775 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 19 | 25 | 44
Weight [Mean (Standard Deviation); unit: Kg] | 15.9 (2.53) | 16.5 (3.87) | 16.2 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation
Description: It is defined as the time from placement of Airtraq or Miller laryngoscope into the mouth till appearance of the capnograph waveform
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 30 | 30
seconds | 15.13 (1.33) | 11.53 (0.49)

2. Secondary Outcome: Number of Intubation in First Attempts;
Description: A single insertion of the Airtraq or a single insertion of the Miller laryngoscope blade into the mouth with passing the endotracheal tube beyond the glottis was considered as an attempt.
Time Frame: 5 minutes
Measure: Number; unit: Intubations
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 30 | 30
Intubations | 25 | 29

3. Secondary Outcome: Ease of Intubation.
Description: The intubating anaesthesiologist graded the ease of intubation for both techniques on a visual analogue scale from 1 to 10, 10 being most difficult or failed intubation and 1 being very easy intubation.
Time Frame: 5 minutes
Measure: Median (Inter-Quartile Range); unit: scores on visual analogue scale
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 30 | 30
scores on visual analogue scale | 5 [3.75 to 6] | 3 [2 to 3.25]

4. Secondary Outcome: Percentage of Glottic Opening Scoring.
Description: The Percentage of glottic opening score represents the percentage of glottic opening seen, defined by the linear span from the anterior commissure to the interarytenoid notch
Time Frame: 5 minutes
Measure: Median (Inter-Quartile Range); unit: percentage of glottic opening
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 30 | 30
percentage of glottic opening | 75 [66 to 100] | 100 [93 to 100]

5. Secondary Outcome: Overall Intubation Success Rate.
Description: It is the number of participants who were successfully intubated after first, second or third attempts. Success of intubation is defined as placement of endotracheal tube inside the trachea, confirmed by bilateral chest auscultation and square wave capnograph tracing.
Time Frame: 5 minutes
Measure: Number; unit: participants
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 30 | 30
participants | 30 | 30

6. Secondary Outcome: Number of Esophageal Intubation.
Description: Insertion of tracheal tube inside the esophagus
Time Frame: 5 minutes
Measure: Number; unit: esophageal intubation
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 30 | 30
esophageal intubation | 4 | 0

7. Secondary Outcome: Number of Participants With Airway Trauma
Description: Airway trauma was defined as blood detected on the blades of laryngoscopes, blood on endotracheal tube after extubation or tongue-lip-dental trauma.
Time Frame: 5 minutes
Measure: Number; unit: participants
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Number analyzed (Participants) | 30 | 30
participants | 3 | 1

ADVERSE EVENTS:
Arm/Group | Intubation With Miller's Blade | Intubation With Airtraq Laryngoscope
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less